CLINICAL TRIAL: NCT01319903
Title: A Single Ascending, Placebo-controlled, Double-blind Study in Healthy Male Subjects to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the New Humanized Monoclonal Antibody CaCP29
Brief Title: Clinical Assessment of Safety and Tolerability of the New Monoclonal Humanized Antibody CaCP29
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IFX-1-P1.1; 2010-023647-15 (EudraCT Number)
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Drug Safety
Keywords: sepsis; inflammation; complement; immune system
MeSH Terms: conditions — Sepsis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: CaCP29, a humanized monoclonal antibody — CaCP29 or placebo single i.v. infusion in ascending doses in healthy human males

SUMMARY:
The novel humanized monoclonal antibody CaCP29 was developed to control the inflammatory response to various stimuli in humans and espacially during sepsis. Purpose of this phase I clinical trial in healthy human males is to investigate various parameters concerning safety and tolerability of CaCP29 and assess pharmacokinetic and pharmacodynamic parameters.

DETAILED DESCRIPTION:
The acute inflammatory innate host response, as being present during the development of sepsis and various other acute inflammatory diseases, represents a powerful mechanisms which can lead to destruction of host tissue and severe organ dysfunction. CaCP29 was developed to lower the complement mediated acute inflammatory response and thereby control the extend of a strongly activated often times self-destructive inflammatory response by controlling activation of a key inflammatory mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Male, Caucasian subjects aged between 18-40 years (inclusive)
* Healthy subjects as determined by medical history, physical examination
* Body weight between 70 - 100 kg and BMI between 19 and 29 kg/m2, extremes incl
* ECG recording based on a 12-lead ECG which is normal (PR < 210 ms, QRS <110 ms, QTC 380 -430 ms) or contains only slight deviations
* Normal vital signs (after 5 minutes resting), blood pressure values (systolic > or equal to 100 and < or equal to 140 mmHg, diastolic > or equal to 50 and < or equal to 90 mmHg), heart rate between 45 and 90 beats per minute (bpm), body temperature < 37.5°C
* Subjects who are able and willing to give written informed consent
* Normal white blood cell count, CRP and IL-6 at screening and Day -1
* Subjects must be using two acceptable methods for contraception (e.g. spermicide and condom) during the study and refrain from fathering a child in the 3 months following dosing

Exclusion Criteria:

* In the opinion of the investigator subjects with clinically significant history or presence of cardiovascular, respiratory, renal, hepatic, metabolic, endocrinological, gastrointestinal, hematological, neurological, dermatological, psychiatric diseases, cancer or other major diseases;
* Infection or known inflammatory process;
* Known autoimmune diseases or immunodeficiency or known family history of autoimmune diseases or immunodeficiency;
* Clinical significant allergic disease;
* Known serum hepatitis or who are carriers of the Hepatitis B surface antigen or Hepatitis C antibodies or with a positive result to the test for HIV 1/2 antibodies;
* Subjects who have received an investigational drug and/or a vaccination within 3 months prior to start of the treatment in study and those who anticipate receipt of a vaccine within 2 months after the last dose of study drug;
* Subjects, who have received prior treatment within 1 year with monoclonal antibodies or other biologic agents;
* The use of any concomitant prescription or non-prescription medication within 14 days prior to the first administration of study medication until follow-up; or treatment with medication that may affect immune function (e.g. immunoglobulins, corticosteroids) within 6 months before dosing;
* Donation of blood (>400 ml) or blood products within the last 3 months prior to admission to the clinical unit or plasmapheresis within 4 weeks prior to study start;
* Definite or suspected personal history of adverse reactions or hypersensitivity to drugs especially to the ingredients of the trial compound or to compounds with a similar structure;
* Use of more than 5 cups or glasses of coffee, tea and / or cola per day;
* Presence or history of drug and/or alcohol abuse or an average daily intake of more than 20 g alcohol per day;
* Positive test for alcohol or drugs at screening and/or on Day -1;
* Smokers of > 5 cigarettes/day or equivalent;
* Subjects who are unlikely to be compliant and attend scheduled clinic visits as required;
* Participation in this study on a previous dose level

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number and extent of changes in safety relevant parameters after injection of CaCP29 | pre-dose, days 1,2,3,7,14,28 and 70
  Safety relevant parameters include changes from baseline of:
  * cytokine levels over time (IL-6, IL-8, IFN-gamma, TNF-alpha, IL-10)
  * CH50 activity over time
  * standard hematology, clinical chemistry and coagulation laboratory parameters
  * 12-lead ECG
  * vital signs

SECONDARY OUTCOMES:
Assessment of pharmacokinetic parameters of CaCP29 over time | pre-dose, day 1,2,3,7, 14, 28 and 70
  * Area under the plasma concentration versus time curve (AUC) of CaCP29
  * Peak Plasma Concentration (Cmax) of CaCP29 and time to reach Cmax
  * terminal phase half-life
  * clearance
  * volume of distribution during the terminal phase
Number of Participants developing anti-CaCP29 antibodies - Immunogenicity | pre-dose, days 28 and 70
Bioactivity of CaCP29 in human whole blood over time after injection | pre-dose, days 1,2,3,7,14,28 and 70

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — FOCUS Clinical Drug Development GmbH Stresemannallee 6 41460 Neuss Germany
Locations (1):
- FOCUS Clinical Drug Development GmbH, Neuss, North Rhine-Westphalia, Germany